CLINICAL TRIAL: NCT04070729
Title: Comparative Evaluation of Local Injectable Platelet Rich Fibrin and Hyaluronic Acid as Adjunctive to Non Surgical Periodontal Therapy: a Randomized Placebo Controlled Clinical Trial
Brief Title: Injectable Platelet Rich Fibrin With Non Surgical Periodontal Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Dental Sciences, Bareilly, Uttar Pradesh, India (Other)
Responsible Party: Principal Investigator, ASHISH AGARWAL, Clinical professor, institute of dental sciences, bareilly, Institute of Dental Sciences, Bareilly, Uttar Pradesh, India
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IEC/IDS50/2019
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: CHRONIC PERIODONTITIS
MeSH Terms: conditions — Chronic Periodontitis | interventions — DBAE cellulose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Negative control (Placebo Comparator): Placebo gel
  Interventions: Other: Placebo gel
- Test group 1 (Experimental): Hyaluronic acid gel
  Interventions: Drug: Hyaluronic acid gel
- Test group 2 (Experimental): injectable prf
  Interventions: Biological: Platelet rich fibrin

INTERVENTIONS:
Other: Placebo gel — Localized subgingival application
  Other Names: Cellulose gel
  Arms: Negative control
Drug: Hyaluronic acid gel — Localized subgingival application
  Arms: Test group 1
Biological: Platelet rich fibrin — Localized subgingival application
  Arms: Test group 2

SUMMARY:
Clinical evaluation of local subgingival application of injectable platelet-rich fibrin ( i-PRF ) for chronic periodntitis as adjunctive to non surgical therapy and compare it with hyaluronic acid.

120 periodontal patients will receive a scaling and root planing ( non surgical periodontal therapy). Equal number of patients will receive subgingival application of i-PRF, hyaluronic acid or placebo gel as the adjunction to non surgical therapy.

DETAILED DESCRIPTION:
The aim of the study is to evaluate and compare the clinical efficacy of subgingival application of i-PRF and hyaluronic acid gel as adjunctive to non-surgical periodontal therapy. 120 periodontal patients will receive traditional mechanical supra and subgingival scaling and root planing. Patients were randomly allocated in three groups. Group 1, 2 and 3 will receive subginigval application of placebo, hyaluronic acid gel and i prf respectively. Clinical parameters will be evaluated: plaque index (PI), gingival index (GI), bleeding on probing (BOP), probing depth (PD), clinical attachment level (CAL), gingival recession (GR). Clinical measurements will be performed at baseline, 1 month and at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients are in general good health.
* Patients having minimum of 20 permanent teeth.
* They have not taken medication known to interfere with periodontal tissue health or healing in the preceding 6 months.
* Presence of periodontal pockets (≥5 mm) and clinicala ttachment level > 5 mm.

Exclusion Criteria:

* Immunosuppressive systemic diseases (like cancer, AIDS, diabetes etc.)
* Clotting and Hematological disorders
* Patients with grade III mobility.
* Patients with smoking and alcohol consuming habit.
* Pregnant and lactating female.
* Medications influence on the gingival and periodontal tissues (like calcium channel blockers, or Long-term steroid use)
* The teeth with poor filling and ill fitted restorations

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-28 (Estimated); Primary Completion 2019-11-28 (Estimated); Study Completion 2020-01-25 (Estimated)

PRIMARY OUTCOMES:
Clinical attachment level (CAL) | 3 Months
  Measure as the change in distance from the cementoenamel junction to the bottom of the gingival sulcus by using a periodontal probe (UNC 15 "University of North Carolina")

SECONDARY OUTCOMES:
Probing pocket depth | 3 Months
  Measure as the change in distance from the gingival margin GM to the bottom of the gingival sulcus by using a periodontal probe (UNC 15 "University of North Carolina")

IPD SHARING:
Plan to Share IPD: No